CLINICAL TRIAL: NCT05845840
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, Single Ascending Dose (SAD) Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BRII-297 in Healthy Adult Subjects
Brief Title: A Study of BRII-297 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brii Biosciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRII-297-001
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-08

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRII-297 (Experimental): Participants will receive a BRII-297 by Intramuscular injection
  Interventions: Drug: BRII-297
- Placebo (Placebo Comparator): Participants will receive placebo by Intramuscular injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BRII-297 — Escalating doses of BRII-297 will be given in different cohorts i.e., Cohorts 1 through 6
  Other Names: Escalating doses of BRII-297
  Arms: BRII-297
Drug: Placebo — Escalating doses of placebo will be given in different cohorts i.e., Cohorts 1 through 6
  Other Names: Placebo to match
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and pharmacokinetics of BRII-297 in healthy adult subjects. The main aim of the study is to evaluate the safety and tolerability after single dose intramuscular administration of BRII-297. The study also aims at characterizing the PK profiles of BRII-297 and brexanolone after single dose intramuscular administration.

Participants will be enrolled in 6 cohorts (3 planned and 3 optional) with 6 participants per cohort [(4 active: 2 placebo) - Cohorts 1 & 2] and 10 participants per cohort [(8 active: 2 placebo) - Cohorts 3 to 6].

Randomization for each cohort will be a two-step process. Sentinel subjects for each cohort will include 2 female subjects randomized 1:1 to BRII-297 or placebo who will be observed for at least 24 hours to ensure no significant safety events before administering study drug to the remaining non-sentinel subjects.

The estimated total duration for each subject is up to 43 days, including screening period (28 days), dosing period (1 day), and post-dose follow-up period (14 days). IM injections will be administered in the gluteal muscle.

Each participant in all cohorts will begin their inpatient stay at the clinical investigational site on Day -1 and remain as an inpatient at the site for sample collection and assessments for 15 days post dose (Day 15). Participants will be released at the end of the inpatient period.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 to 50 years inclusive, at the time of signing informed consent.
2. Capable of giving signed informed consent as described in the protocol which includes compliance with the requirements and restrictions listed in the informed consent and in the protocol in the opinion of the investigator.
3. Subjects who are healthy as determined by medical evaluation including medical history, physical examination, cardiac monitoring using 12-lead ECG, and laboratory tests in the opinion of the investigator.
4. Female or male

   a. Female subjects i. A female subject is eligible to participate if
   * of non-childbearing potential defined as premenarchal, or premenopausal with documented (subject's self-report) bilateral tubal ligation or occlusion, bilateral oophorectomy, bilateral salpingectomy, or hysterectomy; or
   * postmenopausal, documented as 12 months of spontaneous amenorrhea prior to Day 1, and in questionable cases, a blood sample at screening with simultaneous follicle stimulating hormone (FSH) consistent with postmenopausal status (refer to laboratory reference ranges for confirmatory levels); or
   * of childbearing potential, not pregnant, not lactating and agrees to use one of the following acceptable methods of contraception until 30 days after the last dose of study drug:

     * total abstinence from sexual activities, or
     * double barrier method, or
     * an intrauterine device or system, or
     * established use of hormonal contraceptives including oral, implantable, injectable or transdermal contraceptives.

       b. Male subjects i. Male subjects with female partners of childbearing potential must comply withthe following contraception requirements from the time of study drug until90 days after the last dose of study drug administration.
   * total abstinence, or
   * vasectomy with documentation (subject's self-report) of azoospermia 90 days prior to Day 1 (without reversal surgery), or
   * barrier form of contraception (condom), and
   * female partner established user of an intrauterine device/system or hormonal contraceptives including oral, implantable, injectable or transdermal contraceptives.

   ii. Male subjects must also agree not to donate sperm until 90 days after dosing.
5. Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1.
6. Has venous access sufficient to allow for blood sampling.
7. Has a body mass index (BMI) within the range of greater than or equal to 18.0 kg/m2 and less than or equal to 35 kg/m2, and, in the opinion of the investigator, the subject's body habitus would not preclude the ability to correctly inject intramuscularly at the site of injection.
8. Has a maximum body weight of 120 kg.
9. Agrees to abstain from strenuous exercise for 1 week before study Day -1 and during confinement.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, infectious, cardiovascular, gastrointestinal, neoplastic (except for basal or squamous cell cancer), neurological, or psychiatric disorder (as determined by the Investigator) capable of significantly altering the absorption of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of the data.
2. Any major surgical procedure or hospitalization within 6 months prior to Day -1 or during the study, unless deemed not clinically significant by the Investigator.
3. A history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
4. History or presence of an abnormal ECG which, in the Investigator's opinion, is clinically significant. A QTc interval duration Fridericia greater than 450 ms obtained as an average from triplicate screening ECGs after at least 10 minutes rest at screening.
5. Systolic blood pressure greater than 140 mmHg or a diastolic blood pressure of greater than 90 mmHg after approximately 10 minutes rest at screening.
6. Calculated glomerular filtration rate of less than 60 mL/min/1.73m2 by estimated glomerular filtration rate (eGFR) using standardized local clinical methodology.
7. History of alcohol or other substance disorders within 1 year prior to screening, or recent use of drugs of abuse or a positive urine screen for drugs of abuse at screening in the opinion of the Investigator.
8. History of depression or suicidal thoughts and/or behaviors within 1-year prior to screening in the opinion of the Investigator and assessed by S-STS at screening.
9. Has an average weekly alcohol intake that exceeds 10 units per week within 30 days prior to screening. One unit: 1 glass of wine 5 oz or 150 mL; 12 oz or 360 mL of beer; 1.5 oz or 45 mL of distilled spirits.
10. Are unwilling to stop alcohol consumption within 72 hours prior to Day -1 (as confirmed by alcohol breath screen test) and for the duration of the study.
11. Use any tobacco- or nicotine-containing products including, but not limited to cigarettes, electronic cigarettes (of any kind), pipes, vapes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to screen, Day -1 (as confirmed by cotinine testing), and during the study.
12. Positive drug testing at screening and/or at Day -1. Subjects should refrain from eating poppy seed-containing food (e.g., poppy cake) at least 3 days before admission as this can falsify the urine drug screen.
13. History of intolerance to IM injection.
14. Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study.
15. Donated more than 500 mL of blood within 90 days before study drug administration.
16. History of clinically significant chronic liver disease from any cause, presence of hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus antibody.
17. History of hepatic decompensation, including ascites, hepatic encephalopathy and/or esophageal or gastric varices.
18. Positive COVID test on Day -1 (test conducted as per site standard procedures).
19. Is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies (e.g., St. John's wort, milk thistle) or supplement supra-therapeutic doses of vitamins within 14 days (or 5 half-lives, whichever is longer) prior to Day 1 and throughout the study, except for those approved by the Investigator, Medical Monitor, and/or Brii Biosciences.
20. Use of antiplatelet, anticoagulant, or antiepileptic medications within 30 days prior to Day 1 and throughout the study.
21. Use of oral hypoglycemics, diuretics and uricosurics, antidepressants, opioids or centralnervous system acting drugs, such as benzodiazepines, within 14 days before Day 1 andthroughout the study.
22. Consumption of foods or juices containing cranberries or pineapples, Seville oranges,grapefruit, pomegranate or caffeine (xanthine-containing products) within 72 hours priorto Day 1 and throughout the study, unless deemed acceptable by the Investigator.
23. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days or 5 half-lives of the investigational product (whichever is longer).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events receiving BRII-297 compared to placebo | Time Frame: Day 0 - Day 15
  To assess the safety and tolerability of a single infusion of BRII-297 as assessed by frequency of drug related adverse events, graded by severity.
Number of participants with abnormal clinical vital signs | Time Frame: Day 0 - Day 15
  Vital signs include pulse rate, blood pressure, respiratory rate and tympanic temperature
Number of participants with abnormal clinically significant 12-lead electrocardiogram (ECG) readings | Time Frame: Day 0 - Day 15
Number of participants with abnormal clinically significant clinical laboratory results | Time Frame: Day 0 - Day 15
  Clinical laboratory tests include hematology, clinical chemistry, and liver function tests.
Number of participants with abnormal S-STS - Sheehan Suicidality Tracking Scale (self-report) results | Time Frame: Day 1 - Day 15
  Each question is rated from 0 to 4, with the highest score the worse outcome.
Number of participants with abnormal SSS - Stanford Sleepiness Scale (self-report) results | Time Frame: Day 1 - Day 15
  The SSS (self-report) is a subjective measure of sleepiness, The minimum value is 1 (active) and the maximum value is 7 (nearly asleep).
PK of BRII-279 and brexanolone: Maximum observed plasma drug concentration Cmax | Time Frame: Day 0 - Day 15
  The Cmax PK parameter calculated based on the observed plasma drug concentration versus time curve
PK of BRII-279 and brexanolone: Time to maximum observed plasma drug concentration (Tmax) | Time Frame: Day 0 - Day 15
  The PK parameter calculated will be Time to maximum observed plasma drug concentration (Tmax).
PK of BRII-279 and brexanolone: Area under the curve from time 0 to last measurable concentration (AUClast) | Time Frame: Day 0 - Day 15
  The PK parameters calculated will be Area under the plasma drug concentration-time curve from time 0 to last measurable concentration (AUClast).
PK of BRII-279 and brexanolone: Area under the curve from time 0 to infinity (AUC0-inf) | Time Frame: Day 0 - Day 15
  The PK parameters calculated will be Area under the curve from time 0 to infinity (AUC0-inf).
PK of BRII-279 and brexanolone: Terminal elimination half-life (T ½) | Time Frame: Day 0 - Day 15
  The PK parameter of Terminal elimination half-life (T ½) is calculated based on the plasma drug concentration-time curve
PK of BRII-279 and brexanolone: Apparent clearance after extravascular administration (CL/F) | Time Frame: Day 0 - Day 15
PK of BRII-279 and brexanolone: Apparent volume of distribution (Vz/F) | Time Frame: Day 0 - Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Demi Martin, Principal Investigator — CMAX
Locations (1):
- CMAX, Adelaide, South Australia, Australia